CLINICAL TRIAL: NCT06042647
Title: A Demonstration of the Anti-Inflammatory Effects of 0.045% Tazarotene/0.01% Halobetasol Lotion as Compared to 0.05% Clobetasol Propionate Cream in the Treatment of Psoriasis
Brief Title: Anti-Inflammatory Effects of 0.045% Tazarotene/0.01% Halobetasol Lotion in Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dermatology Consulting Services, PLLC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DCS-69-22
Record Dates: First submitted 2023-09-06; First posted 2023-09-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — halobetasol; tazarotene; Clobetasol

STUDY DESIGN:
Intervention Model Description: One product applied to psoriasis on the right side of the body and a second product applied to the left side of the body. The right and left side product applications will be randomized.
Who Masked: Investigator
Masking Description: Investigator will not know which product is applied to the right and left psoriasis target plaque.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.01% Halobetasol and 0.045% Tazarotene Lotion (Active Comparator): 0.01% Halobetasol and 0.045% Tazarotene Lotion (Duobrii)Applied to designated target plaque at bedtime.
  Interventions: Drug: 0.01% Halobetasol; Drug: 0.045% Tazarotene
- Clobetasol Propionate 0.05% Cream (generic) (Active Comparator): Clobetasol Propionate 0.05% Cream (generic)Applied to designated target plaque at bedtime.
  Interventions: Drug: 0.05% Clobetasol Propionate

INTERVENTIONS:
Drug: 0.01% Halobetasol — Drug to be applied at bedtime to designated target psoriasis plaque at bedtime.
  Arms: 0.01% Halobetasol and 0.045% Tazarotene Lotion
Drug: 0.045% Tazarotene — Drug to be applied in combination with 0.01% Halobetasol to the designated psoriasis plaque at bedtime.
  Arms: 0.01% Halobetasol and 0.045% Tazarotene Lotion
Drug: 0.05% Clobetasol Propionate — Drug to be applied to designated psoriatic plaque at bedtime.
  Arms: Clobetasol Propionate 0.05% Cream (generic)

SUMMARY:
The objective of this research is to demonstrate superior anti-inflammatory effects, as demonstrated by a reduction in TNF-a and IL-17A, with tazarotene/halobetasol lotion in patients with mild to moderate plaque type psoriasis as compared to clobetasol propionate 0.05% cream.

DETAILED DESCRIPTION:
Male or female subjects with mild to moderate plaque type psoriasis will present to the research center for evaluation for study entry. They will have been advised to present to the research center with clean skin and no topical products applied to the body, including medications, moisturizers, sunscreens, etc. If found to be suitable by meeting all inclusion criteria and none of the exclusion criteria, subjects will undergo selection of 2 target plaques by the dermatologist investigator. Each plaque will be graded for erythema, scaling, and induration. An Investigational Global Assessment (IGA) score will be assigned for each plaque. Plaques must have an IGA of mild (2) or moderate (3) to qualify for inclusion. The subjects will also assess each plaque for redness, thickness, and scaling. Each of the plaques will be photographed.The subjects will undergo D-squame tape strip removal of each of the 2 target psoriasis plaques. One plaque will serve as the tazarotene/halobetasol lotion treated plaque and the other will serve as the clobetasol propionate 0.05% cream treated plaque. 10 D-squames will be obtained with from each plaque. 5 tape strips will be placed in each glass jar. One jar will contain the even tape strips and the other jar will contain the odd tape strips. 10 D-squames will also be taken from normal skin to serve as a negative control in an individual without psoriasis. 5 tape strips will be placed in each glass jar. One jar will contain the even tape strips and the other jar will contain the odd tape strips. The D-squames will be frozen in a -80C freezer for later assessment. Five tape strips will be analyzed together to obtain adequate material for ELISA analysis. Two specimens jars will be prepared for from each of the 2 target plaques. One jar will be analyzed with the second jar serving as a back up.The subjects will have a number assigned to each of the treatment plaques. The numbers will be recorded on a body map. Two copies will be prepared. One copy will remain at the research center and the second copy will be provided to the subject. Each subject will receive one tube of tazarotene/halobetasol lotion for application to one randomized target plaque and a tube of clobetasol propionate 0.05% cream to apply the second randomized target plaque.Subjects will be provided with a diary. They will be instructed to apply the study product at bedtime to the designated target plaque. Care must be taken to apply the proper product to the proper plaque. Subjects will be instructed to return to the research center in 4 weeks. A reminder text for compliance will be provided prior to the week 4 visit.Subjects will return to the research center at week 4. The dermatologist investigator will evaluate each plaque for erythema, scaling, and induration. An Investigational Global Assessment (IGA) score will be assigned for each plaque. The subjects will also assess each plaque for redness, thickness, and scaling. Each of the plaques will be photographed. The subjects will undergo D-squame tape strip removal of 10 tape strips for each of the 2 target psoriasis plaques. Five tape strips will be placed in each jar with one jar receiving the even tape strips and the other jar receiving the odd tape strips. The D-squames will be frozen in a -80C freezer for later assessment. Subjects will discontinue treatment of the plaques at this time. All medication and study diaries will be collected. Subjects will be asked to return to the research center at week 8. A reminder text for compliance will be sent prior to the week 8 visit.Subjects will return to the research center at week 8. No treatment will be applied to the target plaques for the past 4 weeks. The dermatologist investigator will evaluate each plaque for erythema, scaling, and induration. An Investigational Global Assessment (IGA) score will be assigned for each plaque. The subjects will also assess each plaque for redness, thickness, and scaling. Each of the plaques will be photographed. The subjects will undergo D-squame tape strip removal 10 times for each of the 2 target psoriasis plaques. Five tape strips will be placed in each jar with one jar containing the even tape strips and the other jar containing the odd tape strips. The D-squames will be frozen in a -80C freezer for later assessment. Subjects will complete their study participation at this time.The D-squames will be analyzed using ELISA for the amount of TNF-a and IL-17A present after 4 weeks of treatment with tazarotene/halobetasol lotion to one randomized target plaque and clobetasol propionate 0.05% cream to apply the second randomized target plaque. Treatment will be discontinued at week 4 and subjects will remain untreated for the subsequent 4 weeks. At week 8, D-squames will be analyzed using ELISA for the amount of TNF-a and IL-17A present after 4 weeks off treatment with tazarotene/halobetasol lotion to one randomized target plaque and clobetasol propionate 0.05% cream to apply the second randomized target plaque. This research will allow comparison between a retinoid/topical corticosteroid combination and a topical corticosteroid alone in terms of inflammatory mediator reduction. It will also provide insight into the ability of a retinoid/topical corticosteroid combination to produce longer lasting inflammatory mediator reduction than a topical corticosteroid alone.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant females 18+ years of age.
2. Plaque type mild to moderate psoriasis suitable for topical treatment.
3. The presence of 2 plaques suitable for tape stripping
4. Subjects must be willing to allow a series of tape pieces to be pressed and removed from 2 target psoriasis plaques.
5. Subjects must be in general good health as determined from a medical history.
6. Subjects must read and sign the informed consent form after the nature of the study has been fully explained.

Exclusion Criteria:

1. Subjects with known allergies or sensitivities to ingredients contained in the test products.
2. Subjects with an allergy to latex or adhesives.
3. Subjects with pustular or erythrodermic psoriasis.
4. Subjects who are pregnant or nursing or planning to become pregnant during the course of the study.
5. Subjects who are currently participating in any other clinical study (i.e., dermal patch, use tests, investigational drug or devices, etc.).
6. Subjects viewed by the investigator as not being able to complete the study.
7. Subjects using any type of lotion, medication, or other topical product to the psoriasis plaques.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Concentration of TNF-a and IL-17A in Psoriatic Plaques | 8 weeks
  The primary outcome is to compare the concentration of TNF-a and/or IL-17A after discontinuing treatment for 4 weeks with tazarotene/halobetasol lotion as compared to clobetasol propionate 0.05% cream.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consulting Services, PLLC, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No